CLINICAL TRIAL: NCT02373800
Title: Elastography for Evaluating Cervical Maturity in Preparation for Labor Induction at 37 to 42 Weeks of Gestation
Acronym: ElastoDéclench
Status: Terminated | Type: Observational
Why Stopped: insufficient inclusions
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/VL-02; 2014-A00828-39 (Other: RCB number)
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Labor, Induced
Keywords: Induced; pre-term labor
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population is composed of pregnant women with a medical indication for the induction of pre-term (37-42 weeks of gestation) labor and who are consulting in the participating center.
  Intervention: Cervical ultrasound with elastography
  Interventions: Device: Cervical ultrasound with elastography

INTERVENTIONS:
Device: Cervical ultrasound with elastography — Following routine vaginal exam with determination of Bishop's score, cervical ultrasound with elastography will be used to determine a cervical hardness score varying from 1 to 10. Patients are then hospitalized and labor induced 12 to 48 hours after the elastography.

SUMMARY:
The primary objective of this study is to determine if a cervical hardness score (determined by cervical ultrasound with elastography) can predict delivery mode (vaginal versus cesarian for slow dilatation (more than 2-3h without fetal suffering) regardless of the induction mode (ocytocin alone or with an intravaginal device releasing PGE2).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. To determine composite criteria (combining elastographic, parity and Bishop score information) that predict delivery mode.

B. To determine the prognostic value of elastography as concerns delivery within 24 hours among patients induced via oxytocin with an intravaginal device releasing PGE2 (Bishop score < 6).

C. To determine the prognostic value of elastography as concerns delivery mode (vaginal versus cesarian for slow dilatation (more than 2-3h without fetal suffering))among patients induced via oxytocin alone.

D. To evaluate the intra- and inter-operator reproducibility of the cervical hardness score determined via elastography.

E. To evaluate the economic impact of using the cervical hardness score from the point of view of the French social system (French health insurance) and the hospital.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Pregnant woman with a medical indication for pre-term labor induction: 37 to 42 weeks of gestation.

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* History of cervical surgery
* Malformation of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of pregnant women with a medical indication for the induction of pre-term (37-42 weeks of gestation) labor and who are consulting in the participating center.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Cervical hardness score | Day 0 (baseline)
  A score varying from 0 to 10 determined during cervical ultrasound with elastography.
Mode of delivery: vaginal delivery versus cesarean | Day 2

SECONDARY OUTCOMES:
Bishop score | Day 0 (baseline)
Parity | Day 0 (baseline)
Time lapsed between labor induction and delivery | Day 2
Induction mode | Day 0 (baseline)
  oxytocin alone or with an intravaginal device releasing PGE2
Cervical hardness score for reproductibility 1 | Day 0 (baseline)
  Second reading (by the same, original operator) of ultrasound+elastography recording
Cervical hardness score for reproductibility 2 | Day 0 (baseline)
  Third reading (by a second operator) of ultrasound+elastography recording
Cost of hospital stay | Expected average of 4-5 days

OTHER OUTCOMES:
Age in years | Day 0 (baseline)
Body mass index | Day 0 (baseline)
Number of previous vaginal deliveries | Day 0 (baseline)
Duration of labor | Day 2
Birthweight of the newborn | Day 2
Maternal complications | Day 2
Complications for the newborn | Day 2
Indication for cesarian: fetal cause, cervical cause, non descent | Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France